CLINICAL TRIAL: NCT00334581
Title: A Study of Irbesartan 150mg Verses 300mg in Chinese Hypertensive Patients With Diabetes and Microalbuminuria
Brief Title: Irbesartan in Chinese Hypertensive Diabetics With Microalbuminuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBES_L_00907
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

ARMS (2):
- 1 (Experimental): Irbesartan 150mg
  Interventions: Drug: Irbesartan
- 2 (Experimental): Irbesartan 300mg
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan — Administration throughout the study period
  Arms: 1
Drug: Irbesartan — Administration throughout the study period
  Arms: 2

SUMMARY:
Primary objective:

* To determine if irbesartan 300mg is better than 150mg in protecting the kidneys in hypertensive patients with diabetes and microalbuminuria.

Secondary objectives:

* To determine how well irbesartan 300mg is tolerated versus 150mg
* To determine the percentage of patients reaching the blood pressure target of 130/80 mmHg

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients, treated or untreated, with type 2 diabetes and urinary albumin excretion rate 20-200ug/min.
* Blood pressure of < 180/110mmHg at baseline
* Normal serum creatinine

Exclusion Criteria:

* Type 1 diabetes
* Use of angiotensin converting enzyme inhibitors or angiotensin receptor blockers in the 5 weeks before recruitment
* Pregnant or lactating women
* Severe hypertension
* Overt nephropathy
* Allergy to study drug

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The difference of urinary albumin excretion rate change | at week 24

SECONDARY OUTCOMES:
Percentage of patients reaching target BP of 130/80mmHg | At week 24
Adverse events | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Jolain, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China